CLINICAL TRIAL: NCT01911949
Title: An Ultrasound Guided Fascia Iliaca Block Placed at the Level of the Inguinal Ligament for Analgesia After Hip Arthroplasty
Brief Title: USFIB at the Inguinal Ligament for Total Hip Arthroplasty
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: McMaster University (Other)
Collaborators: St. Joseph's Healthcare Hamilton (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 12-3688
Record Dates: First submitted 2013-07-26; First posted 2013-07-30 (Estimated); Last update posted 2018-03-22 (Actual); Status verified 2018-03

CONDITIONS: Post Surgical Pain
Keywords: femoral nerve block; ultrasound guided; total hip arthroplasty
MeSH Terms: conditions — Pain, Postoperative | interventions — Bupivacaine; Epinephrine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Single shot femoral nerve block (Experimental): Ultrasound guided Femoral Nerve Block-40ml of bupivacaine 0.5% with epinephrine
  Interventions: Drug: Single shot femoral nerve block
- Placebo femoral nerve block (Placebo Comparator): Sterile normal saline solution
  Interventions: Drug: Single shot femoral nerve block

INTERVENTIONS:
Drug: Single shot femoral nerve block — Nerve block in lingual crease using ultrasound guidance
  Other Names: Femoral Nerve Block with 40ml bupivacaine plus 0.5% epinephrine

SUMMARY:
Hip replacement surgery is one of the most common elective surgeries in Canada and with this surgery, there is considerable pain after the operation. By decreasing the amount of pain after surgery, the patients may be able to move and walk quicker, resulting in easier physiotherapy sessions, shorter hospital stays and may help to avoid adverse outcomes like nausea and vomiting and being overly sedated. By using ultrasound guided femoral nerve block, it may be an alternative for pain management with minimal side effects for patients having hip replacement surgery.

DETAILED DESCRIPTION:
Ultrasound guided femoral blocks have been studied since the late 90's. A study published in 1997 by Marhofer et al. pointed that ultrasound guidance in a 3-in-1 block (femoral, obturator, lateral cutaneous nerves), improved the quality of the sensory block and reduced the onset time when compared with a nerve-stimulation technique in patients undergoing hip surgery after trauma.(13) In a meta-analysis comparing ultrasound guidance versus electrical nerve-stimulation for peripheral nerve blocks, the authors reported a decreased risk of block failure, shorter procedure time and faster onset time when ultrasound is used.(14)

A systematic review studying the outcomes after Total Hip Arthroplasty concluded that when compared with systemic analgesia the use of femoral nerve block was on unclear benefit.(15) Separate analysis of the two studies included showed that in the Biboulet study, ultrasound was not used to perform the blocks, and pain with activity was not evaluated in the first 24 hours after surgery, time in which the maximum benefit of blocks is observed.(16) In the second study by Singelyn et al. with continuous femoral nerve block, the authors found similar pain relief than with IV Patient Controlled Analgesia morphine with fewer side effects.(17)

While recent publications have demonstrated the analgesia effectiveness of femoral nerve block and fascia iliaca block for hip fractures,(18) there are not references in the literature analyzing the effectiveness of a single shot, ultrasound-guided, femoral nerve block in primary hip arthroplasty. This fact opens up the possibility to continue researching the analgesic effectiveness of this block in a population where the options for handling postoperative pain are limited widely for its side effects together with the use of anticoagulant and anti-thrombotic therapy.

This technique is considered a simple procedure, easy to teach and to learn. If our study shows improvement of the outcomes, it will feasible to incorporate this block as an alternative for pain management after primary hip arthroplasty.

Given the complexity of this proposed randomized-controlled trial, a pilot study was deemed necessary to find out the feasibility and safety of the intervention, rate of patient recruitment and needs for additional personnel.

ELIGIBILITY:
Inclusion Criteria:

1. Patients 18 years or older undergoing unilateral hip arthroplasty.
2. Patient capable to complete informed consent.

Exclusion Criteria:

1. Pediatric population.
2. Inability to complete informed consent.
3. Patient refusal.
4. Contraindication for regional anesthesia: coagulopathy, anticoagulant use, bleeding disorders, local or systemic infection, local anesthesia allergy.
5. Presence of neuromuscular deficit including diabetic peripheral neuropathy.

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 24 (Actual)
Dates: Start 2017-01 (Actual); Primary Completion 2017-08 (Actual); Study Completion 2017-08 (Actual)

PRIMARY OUTCOMES:
The primary outcome is number of patients recruited per week and we hope to recruit 2 patients per week. | Three months

SECONDARY OUTCOMES:
Number of eligible patients consenting to participate. | Three months
Number of patients participating that were randomized and received the study intervention. | Three months
Completion of study data collection forms | Three months
Incidence of respiratory depression and seizures in participating subjects | Three months

CONTACTS AND LOCATIONS:
Overall Officials: Mauricio Forero, MD, Principal Investigator — St. Joseph's Healthcare Hamilton
Locations (1):
- St. Joseph's Heathcare Hamilton, Hamilton, Ontario, Canada

REFERENCES:
- [Background] Rothwell MP, Pearson D, Hunter JD, Mitchell PA, Graham-Woollard T, Goodwin L, Dunn G. Oral oxycodone offers equivalent analgesia to intravenous patient-controlled analgesia after total hip replacement: a randomized, single-centre, non-blinded, non-inferiority study. Br J Anaesth. 2011 Jun;106(6):865-72. doi: 10.1093/bja/aer084. Epub 2011 Apr 13. PMID 21490024